CLINICAL TRIAL: NCT03391154
Title: Efficacy of Low Dose Levothyroxine During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: asu maternity hosp
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Euthyroid Females
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- levothyroxine (Active Comparator): 100 pregnant female with TSH of> 2.5 mU/L but less than 4 mU/L after biochemical diagnosis of pregnancy will receive 50 ug of levothyroxine (eltroxin 50) aspen,Egypt throughout the pregnancy
  Interventions: Drug: levothyroxin
- control (No Intervention): 100 pregnant female with TSH of> 2.5 mU/L but less than 4 mU/L after biochemical diagnosis of pregnancy will not receive any drug throughout the pregnancy

INTERVENTIONS:
Drug: levothyroxin — 90 female received levothroxine
  Arms: levothyroxine

SUMMARY:
the effect using low dose levo thyroxine in pregnant females with TSH level more than 2.5 mU/L in the first trimester on pregnancy outcome

DETAILED DESCRIPTION:
the study aim to detect the effect of low dose levothyroxine 50 ug on pregnant females and compare it with others receiving placebo

ELIGIBILITY:
Inclusion Criteria:

* females with TSH more than 2.5 mU/L and less than 4 mU/L after biochemical diagnosis of pregnancy.

Exclusion Criteria:

* associated endocrinopathies (PCO/ DM/ hyperprolactinemia )
* associated medical condition (HTN/ chronic kidney disease.
* history of recurrent pregnancy loss

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
1st trimester miscarriage | during 1st 13 weeks of pregnancy
  1st trimester spontaneous or missed abortion

SECONDARY OUTCOMES:
adverse pregnancy outcome | last 26 week of gestation
  2nd trimesteric missed or spontaneous abortion ,gestational hypertension,preeclampsia, anemia, abruptio placenta premature delivery , fetal growth restriction, low birth weight

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided